CLINICAL TRIAL: NCT02990936
Title: Prognostic Impact of Tumor Growth Velocity in Head and Neck Squamous Cell Carcinoma Treated by Radio(Chemo)Therapy
Acronym: TGV-PI
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Sponsor
Other Study IDs: TGV-PI01
Record Dates: First submitted 2015-05-28; First posted 2016-12-13 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Tumor Growth
Keywords: hea and neck squamous cell carcinoma; tumor growth; predictive markers; tumoral kinetics
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oropharynx biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- head and neck squamous cell carcinoma: Patients with T1 to T4 head and neck squamous cell carcinoma from oral cavity, oropharynx, larynx and hypopharynx eligible for radiotherapy or concomitant chemoradiotherapy
  Interventions: Other: Tumor delineation

INTERVENTIONS:
Other: Tumor delineation — Measurement of tumor volume and neck nodes volume on a diagnostic CT and a pre-treatment CT by computerized delineation in order to calculate tumor growth velocity and tumor doubling time and describe tumoral kinetics patterns

SUMMARY:
The purpose of this study is to determine the impact of tumor growth velocity on the survival of patients with hea and neck squamous cell carcinoma treated by (chemo-)radiotherapy.

Patients with stages I to IV oropharyngeal primary squamous cell carcinoma (OPSCC) elected for radiotherapy or radiochemotherapy with curative intent will be selected. Tumor volume and number and size of pathological neck lymph nodes (small diameter > 1 cm) will be assessed on diagnostic CT-scan (DiCT) and treatment planning CT-scan (RtCT) using the summation of areas technique. Tumor progression and tumor doubling time will be calculated based on DiCT and RtCT. Tumor proliferation will be assessed on biopsy specimens by Ki67 immunohistochemistry and mitotic index. HPV status will be evaluated by PCR and p16 immunohistochemistry. Ulcerative or exophytic aspect will be noticed. Tumoral kinetics patterns will be correlated with disease free survival and overall survival of patients with HNSCC. These patterns will be compared to HPV status and proliferation markers in order to study their clinical signification [time frame: 5 years] and develop predictive markers of tumor progression for head and neck cancers.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) represents more than 90 percent of head and neck tumors and is one of the most frequent human neoplasms. During the last decades, radiotherapy has emerged as a standard treatment of HNSCC and the number of patients treated with this modality has continuously increased. Moreover, treatment schedules for radiotherapy have improved and require more preparation and are therefore more time consuming. Thus, waiting time prior to radiotherapy becomes a major concern in many countries with reported delays of 70 days or even more.Clinicians involved in treating HNSCC face the problem of rapidly growing tumors but despite significant progress in the understanding of these tumors, their development and progression remain currently unpredictible at the time of diagnosis. In a retrospective trial, Laccourreye et al. studied the time of progression of symptoms and signs (TPSS) before diagnosis and treatment in 966 HNSCC cases and showed that for a given tumor stage, the longer was the TPSS, the better were the vital prognosis, the local and lymph node control. But there is no clear definition of fast growing tumor, with objective measurement.

A CT-scan is perfomed at the time of diagnosis. Several weeks later, a second CT-scan is necessary for treatment planning in order to define the tumoral target volume. This necessity provides the opportunity to compare tumoral volumes on both exams, and thus to assess tumoral progression. In a pilot study conducted with Institut Gustave Roussy, the investigators studied retrospectively the tumor and loco-regional progression in the waiting time between diagnostic and treatment planning CT-scans in a cohort of patients with oropharyngeal squamous cell carcinoma, treated by radio(chemo)therapy between April 2005 and April 2007. The study demonstrated that 53% of the patients presented a tumoral progression of > 50% within a mean waiting time of 42.1 +/- 15.7 days. The investigators consider this situation as regrettable, and prospective trials are clearly needed to determine clinical consequences of these findings.

The current project aims to study prospectively the loco-regional tumoral progression within the waiting time between diagnostic and treatment planning CT-scans in a cohort of patients with OPSCC. Patients with oropharyngeal primary squamous cell carcinoma elected for radiotherapy or radiochemotherapy with curative intent will be selected. Tumor volume, number and size of pathological cervical lymph nodes (small diameter > 1 cm) will be assessed on diagnostic CT-scan (DiCT) and treatment planning CT-scan (RtCT) using the summation of areas technique (computerized delineation). Tumoral progression and tumor doubling time will be calculated based on DiCT and RtCT in order to define different tumoral kinetics patterns. Human papillomavirus (HPV) status will be assessed by polymerase chain reaction (PCR) and p16 immunohistochemistry. As primary objective, the investigators will study the tumoral kinetics patterns with disease free survival (DFS) and overall survival (OS) in patients with OPSCC in order to study their clinical signification [time frame: 5 years]. As secondary objectives, the investigators will correlate the tumoral kinetics patterns with HPV status of patients with OPSCC, and compare tumoural kinetics to proliferation markers (Ki67, mitotic index) in order to develop predictive markers of tumour progression for head and neck cancers. An other complementary objective will compare tumor kinetics patterns with endoscopic aspect (ulcerative versus exophytic)

ELIGIBILITY:
Inclusion Criteria:

* clinical and anatomopathological diagnosis of a head and neck squamous cell carcinoma (T1 to T4) (oral cavity, oropharynx, larynx, hypopharynx)
* multidisciplinary decision for radiotherapy or concomitant radiochemotherapy eligibility

Exclusion Criteria:

* metastatic disease
* primary surgical management
* contraindications to iodine contrast injection: anaphylaxis and renal insufficiency
* tumor not visible on CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All T1 to T4 patients under eligibility criteria with head and neck squamous cell carcinoma admitted to the investigators' tertiary centers will be selected.
  Centre hospitalier Universitaire Godinne is a belgian provincial tertiary center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years follow-up after recruitment
disease-free survival | 5 years

SECONDARY OUTCOMES:
correlation between kinetics patterns and HPV status | 5y follow-up

OTHER OUTCOMES:
correlation between kinetics patterns and proliferation markers | 5y follow-up
correlation between kinetics patterns and endoscopic aspect of the tumor | 5y follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Van der Vorst, MD, PhD, Principal Investigator — CHU Dinant Godinne
Locations (2):
- Belgium (2):
  - Clinique Ste-Elisabeth, Namur
  - CHU Dinant Godinne, Yvoir

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Waaijer A, Terhaard CH, Dehnad H, Hordijk GJ, van Leeuwen MS, Raaymakers CP, Lagendijk JJ. Waiting times for radiotherapy: consequences of volume increase for the TCP in oropharyngeal carcinoma. Radiother Oncol. 2003 Mar;66(3):271-6. doi: 10.1016/s0167-8140(03)00036-7. PMID 12742266
- [Background] Jensen AR, Nellemann HM, Overgaard J. Tumor progression in waiting time for radiotherapy in head and neck cancer. Radiother Oncol. 2007 Jul;84(1):5-10. doi: 10.1016/j.radonc.2007.04.001. Epub 2007 May 9. PMID 17493700
- [Background] Brouha XD, Op De Coul B, Terhaard CH, Hordijk GJ. Does waiting time for radiotherapy affect local control of T1N0M0 glottic laryngeal carcinoma? Clin Otolaryngol Allied Sci. 2000 Jun;25(3):215-8. doi: 10.1046/j.1365-2273.2000.00347.x. PMID 10944052
- [Background] De Meerleer GO, Vakaet LA, De Gersem WR, De Wagter C, De Naeyer B, De Neve W. Radiotherapy of prostate cancer with or without intensity modulated beams: a planning comparison. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):639-48. doi: 10.1016/s0360-3016(00)00419-3. PMID 10837946
- [Background] Mackillop WJ, Zhou Y, Quirt CF. A comparison of delays in the treatment of cancer with radiation in Canada and the United States. Int J Radiat Oncol Biol Phys. 1995 May 15;32(2):531-9. doi: 10.1016/0360-3016(94)00662-5. PMID 7751195
- [Background] O'Rourke N, Edwards R. Lung cancer treatment waiting times and tumour growth. Clin Oncol (R Coll Radiol). 2000;12(3):141-4. doi: 10.1053/clon.2000.9139. PMID 10942328
- [Background] Primdahl H, Nielsen AL, Larsen S, Andersen E, Ipsen M, Lajer C, Vestermark LW, Andersen LJ, Hansen HS, Overgaard M, Overgaard J, Grau C; DAHANCA. Changes from 1992 to 2002 in the pretreatment delay for patients with squamous cell carcinoma of larynx or pharynx: a Danish nationwide survey from DAHANCA. Acta Oncol. 2006;45(2):156-61. doi: 10.1080/02841860500423948. PMID 16546860
- [Background] Robinson D, Massey T, Davies E, Jack RH, Sehgal A, Moller H. Waiting times for radiotherapy: variation over time and between cancer networks in southeast England. Br J Cancer. 2005 Apr 11;92(7):1201-8. doi: 10.1038/sj.bjc.6602463. PMID 15785752